CLINICAL TRIAL: NCT01140529
Title: A Prospective, Multi-centre, Randomised, Double-blind, Placebo-controlled Comparison of Intravenous Dexmedetomidine and Haloperidol in Treatment of Psychomotor Confusion After Heart Surgery
Brief Title: Dexmedetomidine for the Treatment of Delirium After Heart Surgery
Acronym: DexinDelir
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Thorax-Kärlkliniken (Other)
Responsible Party: Principal Investigator, Sten Walther, Dr, Thorax-Kärlkliniken
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3005099
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative; Delirium; Psychomotor; Confusion
Keywords: Dexmedetomidine
MeSH Terms: conditions — Delirium; Confusion | interventions — Dexmedetomidine; Haloperidol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Haloperidol (Active Comparator)
  Interventions: Drug: Haloperidol
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Bolus and continuous infusion
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Haloperidol — Bolus doses
  Other Names: Haldol
  Arms: Haloperidol
Drug: Saline — Bolus and continuous infusion
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
Primary hypothesis: Dexmedetomidine is equal or superior to haloperidol and placebo in the treatment of psychomotor confusion in patients who are recovering from heart surgery.

Study design:

Multi-centre, prospective, randomised, placebo-controlled double-blind study of dexmedetomidine vs. haloperidol for treatment of psychomotor confusion after cardiac surgery. Data will be analyzed in two steps: The primary comparison is between placebo and dexmedetomidine. If the effect of dexmedetomidine is significant, a secondary comparison between dexmedetomidine and haloperidol will follow.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Clinical need for treatment of psychomotor confusion unresponsive to standard analgesic medication (RASS +2 to +3)
* Heart surgery and extracorporeal circulation (ECC) within 7 days
* Written informed consent obtained before surgery
* Mentally competent at the time of written informed consent

Exclusion Criteria:

* Ongoing neuroleptic, propofol and α2 agonist medication
* Intubated patient
* Uncompensated acute circulatory failure at time of randomisation (severe hypotension with mean arterial pressure < 55 mmHg despite volume, vasopressors and IABP)
* Severe bradycardia without pacemaker backup (heart rate < 50 beats/min)
* AV-conduction block II-III (without pacemaker backup)
* Severe hepatic impairment (Serum bilirubin > 101 µmol/l)
* Lithium therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Need for rescue medication | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sten M Walther, MD PhD, Principal Investigator — ThoraxKärlkliniken, University Hospital, Linköping, Sweden
Locations (1):
- ThoraxKärlkliniken, Universitetssjukhuset, Linköping, Sweden